CLINICAL TRIAL: NCT03953651
Title: Clinical Presentation and Outcomes in Patients at Risk of Type II Myocardial InfarctioN in the emerGency Department.
Acronym: COMING
Status: Completed | Type: Observational
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 69HCL18_0913; 2019-A00177-50 (Other: ID-RCB)
Record Dates: First submitted 2019-05-15; First posted 2019-05-16 (Actual); Last update posted 2020-07-28 (Actual); Status verified 2020-07

CONDITIONS: Myocardial Oxygenation Imbalance; Myocardial Infarction
MeSH Terms: conditions — Myocardial Infarction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Patients admitted in the emergency department presenting a myocardial oxygenation imbalance and are therefore at risk for Myocardial Infarction (MI) type 2.
  Interventions: Other: Follow-up

INTERVENTIONS:
Other: Follow-up — Onset of Major Adverse Cardiovascular Event of death from all causes will be collected at 3 and 6 months after inclusion.

SUMMARY:
Type 2 myocardial infarction has been reported in the Universal Definition of Myocardial Infarction for more than 10 years and most studies resulted in a high mortality rate. However, little to nothing is known for both criteria to define myocardial oxygenation imbalance threshold and the outcome of these patients presenting with myocardial oxygenation imbalance.

The aim of this study is to compare the outcome at 6 months for patients admitted in the emergency department with a myocardial oxygenation imbalance, depending on whether a type 2 myocardial infarction occured or not.

ELIGIBILITY:
Inclusion Criteria:

* age 18 years old or older ;
* At least one condition of myocardial oxygenation imbalance :

  * Oxygen saturation below 90% ;
  * Haemoglobin level below 130 grams/Liter (g/L) for men, 120 g/L for women ;
  * Persistent heart rate over 110 beats per minute, for more than 20 minutes ;
  * Persistent systolic blood pressure below 90 millimeters of mercury (mmHg) for more than 20 minutes despite fluid resuscitation ;
  * Persistent systolic blood pressure over 180 mmHg for more than 20 minutes.

Exclusion Criteria:

* Patient admitted with type 1 myocardial infarction ;
* Patient presenting a condition for Non Ischemic Myocardial Infarction (pulmonary embolism, acute stroke, acute kidney failure, etc…)
* Patient who declines to participate;
* Pregnant or breastfeeding women ;
* Patient deprived of liberty (inmate, administrative protection)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female patients at least 18 years old admitted to the emergency department with a myocardial oxygenation imbalance
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2019-07-10 (Actual); Primary Completion 2020-07-09 (Actual); Study Completion 2020-07-09 (Actual)

PRIMARY OUTCOMES:
Onset of a Major Adverse Cardiovascular Event at 6 months | 6 months
  Onset of a Major Adverse Cardiovascular Event such as:
  * Cardiovascular death
  * Non fatal myocardial infarction
  * Admission for acute heart failure
  * Non fatal stroke

CONTACTS AND LOCATIONS:
Overall Officials: Laurent JACQUIN, Dr, Principal Investigator — Hospices Civils de Lyon
Locations (1):
- Hôpital Edouard Herriot, Lyon, France